CLINICAL TRIAL: NCT04684238
Title: A Randomised Active-controlled Study to Compare Efficacy & Safety of Inhaled Isoflurane Delivered by the AnaConDa-S (Anaesthetic Conserving Device) vs IV Midazolam for Sedation in Mechanically Ventilated Paediatric Patients 3-17 Years Old
Brief Title: Effect & Safety of Inhaled Isoflurane vs IV Midazolam for Sedation in Mechanically Ventilated Children 3-17 Years Old
Acronym: IsoCOMFORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sedana Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SED002
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sedation
Keywords: sedation; isoflurane; mechanically ventilation; pediatric; midazolam
MeSH Terms: interventions — Midazolam; Isoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Midazolam (Active Comparator): Midazolam for sedation in the ICU
  Interventions: Drug: Midazolam
- Drug: Isoflurane (Experimental): Volatile for sedation in the ICU
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Midazolam — Solution for Injection/Infusion
  Arms: Drug: Midazolam
Drug: Isoflurane — Inhalation vapour, liquid. Isoflurane delivered by the AnaConDa-S (Anaesthetic Conserving Device)
  Arms: Drug: Isoflurane

SUMMARY:
This is a study to compare safety and efficacy of inhaled isoflurane delivered by the AnaConDa-S (Anaesthetic Conserving Device (ACD)) versus intravenous midazolam for sedation in mechanically ventilated children admitted to an intensive care unit.

DETAILED DESCRIPTION:
This is a phase III, multi-centre, prospective, randomized, active-controlled, assessor-blind study. Primary endpoint: percentage of time of adequately maintained sedation, in absence of rescue sedation, within the COMFORT-B interval (light, moderate, or deep sedation) prescribed at randomization, monitored every 2 hours for an expected minimum of 12 hours (up to 48 hours).

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 3 years to 17 (less than 18) years at the time of randomization, admitted to an ICU/with planned ICU admission.
* Expected mechanical (invasive) ventilation and sedation for at least 12 hours.
* Informed consent obtained from the patient, patient's legal guardian(s)

Exclusion Criteria:

* Ongoing seizures requiring acute treatment.
* Continuous sedation for more than 72 hours at time of randomization.
* Less than 24 hours post cardiopulmonary resuscitation.
* Uncompensated circulatory shock.
* Known or suspected genetic susceptibility to malignant hyperthermia.
* Patients with acute asthma or obstructive lung disease symptoms requiring treatment at inclusion.
* Patient with tidal volume below 30 mL or above 800 mL.
* Inability to perform reliable COMFORT-B assessment in the opinion of the Investigator
* Patients with intracranial pressure (ICP) monitoring or with suspected increase in ICP
* Patients with treatment-induced whole-body hypothermia.
* Patients with pheochromocytoma.
* Patients with prolonged QT interval or with significant risk for prolonged QT interval.
* Patient not expected to survive next 48 hours or not committed to full medical care.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sackey, MD, PhD, Study Director — Sedana Medical
Locations (24):
- France (6):
  - Hôpital Femme-Mère-Enfant Groupe Hospitalier Est, Lyon
  - CHU de NANTES, Hôpital Mère-Enfant, Nantes
  - Hôpital Robert-Debré AP-HP, Paris
  - Hôpitaux Universitaires Paris Sud Site Bicetre, Paris
  - Centre Hospitalier Universitaire de Reims, Reims
  - Hôpitaux Universitaires de Strasbourg Hôpital de Hautepierre, Strasbourg
- Germany (4):
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitätsklinikum Jena, Jena
- Spain (9):
  - Hospital Materno Infantil Sant Joan de Deu Hospital, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Infantil Universitario Niño Jesús Pediatric Intensive Care Unit, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario, Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocio de Sevilla, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Karolinska Universitetssjukhus Solna, Solna, Sweden
- United Kingdom (4):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Imperial College Healthcare NHS Trust, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eifinger F, Hunseler C, Roth B, Vierzig A, Oberthuer A, Mehler K, Kribs A, Menzel C, Trieschmann U. Observations on the effects of inhaled isoflurane in long-term sedation of critically Ill children using a modified AnaConDa(c)-system. Klin Padiatr. 2013 Jul;225(4):206-11. doi: 10.1055/s-0033-1345173. Epub 2013 Jun 24. PMID 23797368
- [Background] Ariyama J, Hayashida M, Shibata K, Sugimoto Y, Imanishi H, O-oi Y, Kitamura A. Risk factors for the development of reversible psychomotor dysfunction following prolonged isoflurane inhalation in the general intensive care unit. J Clin Anesth. 2009 Dec;21(8):567-73. doi: 10.1016/j.jclinane.2009.01.011. PMID 20122588
- [Background] Grant MJ, Balas MC, Curley MA; RESTORE Investigative Team. Defining sedation-related adverse events in the pediatric intensive care unit. Heart Lung. 2013 May-Jun;42(3):171-6. doi: 10.1016/j.hrtlng.2013.02.004. PMID 23643411
- [Background] Hoemberg M, Vierzig A, Roth B, Eifinger F. Plasma fluoride concentrations during prolonged administration of isoflurane to a pediatric patient requiring renal replacement therapy. Paediatr Anaesth. 2012 Apr;22(4):412-3. doi: 10.1111/j.1460-9592.2012.03814.x. No abstract available. PMID 22380747
- [Background] Kruessell MA, Udink ten Cate FE, Kraus AJ, Roth B, Trieschmann U. Use of propofol in pediatric intensive care units: a national survey in Germany. Pediatr Crit Care Med. 2012 May;13(3):e150-4. doi: 10.1097/PCC.0b013e3182388a95. PMID 22079951
- [Background] Kudchadkar SR, Yaster M, Punjabi NM. Sedation, sleep promotion, and delirium screening practices in the care of mechanically ventilated children: a wake-up call for the pediatric critical care community*. Crit Care Med. 2014 Jul;42(7):1592-600. doi: 10.1097/CCM.0000000000000326. PMID 24717461
- [Background] Nolent P, Laudenbach V. [Sedation and analgesia in the paediatric intensive care unit]. Ann Fr Anesth Reanim. 2008 Jul-Aug;27(7-8):623-32. doi: 10.1016/j.annfar.2008.04.014. Epub 2008 Jul 9. French. PMID 18614330
- [Background] Meiser A, Laubenthal H. Inhalational anaesthetics in the ICU: theory and practice of inhalational sedation in the ICU, economics, risk-benefit. Best Pract Res Clin Anaesthesiol. 2005 Sep;19(3):523-38. doi: 10.1016/j.bpa.2005.02.006. PMID 16013698
- [Background] Meyburg J, Dill ML, von Haken R, Picardi S, Westhoff JH, Silver G, Traube C. Risk Factors for the Development of Postoperative Delirium in Pediatric Intensive Care Patients. Pediatr Crit Care Med. 2018 Oct;19(10):e514-e521. doi: 10.1097/PCC.0000000000001681. PMID 30059477
- [Background] Mody K, Kaur S, Mauer EA, Gerber LM, Greenwald BM, Silver G, Traube C. Benzodiazepines and Development of Delirium in Critically Ill Children: Estimating the Causal Effect. Crit Care Med. 2018 Sep;46(9):1486-1491. doi: 10.1097/CCM.0000000000003194. PMID 29727363
- [Background] Playfor S, Jenkins I, Boyles C, Choonara I, Davies G, Haywood T, Hinson G, Mayer A, Morton N, Ralph T, Wolf A; United Kingdom Paediatric Intensive Care Society Sedation; Analgesia and Neuromuscular Blockade Working Group. Consensus guidelines on sedation and analgesia in critically ill children. Intensive Care Med. 2006 Aug;32(8):1125-36. doi: 10.1007/s00134-006-0190-x. Epub 2006 May 13. PMID 16699772
- [Background] Sackey PV, Martling CR, Granath F, Radell PJ. Prolonged isoflurane sedation of intensive care unit patients with the Anesthetic Conserving Device. Crit Care Med. 2004 Nov;32(11):2241-6. doi: 10.1097/01.ccm.0000145951.76082.77. PMID 15640636
- [Background] Sackey PV, Martling CR, Radell PJ. Three cases of PICU sedation with isoflurane delivered by the 'AnaConDa'. Paediatr Anaesth. 2005 Oct;15(10):879-85. doi: 10.1111/j.1460-9592.2005.01704.x. PMID 16176317
- [Background] Tobias JD. Tolerance, withdrawal, and physical dependency after long-term sedation and analgesia of children in the pediatric intensive care unit. Crit Care Med. 2000 Jun;28(6):2122-32. doi: 10.1097/00003246-200006000-00079. PMID 10890677
- [Background] Vet NJ, Ista E, de Wildt SN, van Dijk M, Tibboel D, de Hoog M. Optimal sedation in pediatric intensive care patients: a systematic review. Intensive Care Med. 2013 Sep;39(9):1524-34. doi: 10.1007/s00134-013-2971-3. Epub 2013 Jun 19. PMID 23778830
- [Derived] Miatello J, Palacios-Cuesta A, Radell P, Oberthuer A, Playfor S, Amores-Hernandez I, Barreault S, Biedermann R, Charlo Molina MT, Encarnacion Martinez J, Kuehne B, Mencia S, Mendez MD, Menzel C, Morin L, Oviedo L, Piloquet JE, Falkenhav M, Sackey P, Trieschmann U, Tissieres P; IsoCOMFORT Study Group. Inhaled isoflurane for sedation of mechanically ventilated children in intensive care (IsoCOMFORT): a multicentre, randomised, active-control, assessor-masked, non-inferiority phase 3 trial. Lancet Respir Med. 2025 Oct;13(10):897-910. doi: 10.1016/S2213-2600(25)00203-6. Epub 2025 Jul 15. PMID 40680761

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 patients were randomised in total, 2 patients randomised to isoflurane did not receive treatment and 3 patients receiving treatment did not complete (1 patient receiving isoflurane and 2 patients receiving midazolam)
Groups:
- Drug: Isoflurane: Volatile for sedation in the ICU
  Isoflurane: Inhalation vapour, liquid. Isoflurane delivered by the Anaesthetic Conserving Device (ACD), i.e., Sedaconda ACD-S.
Period: Overall Study
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Started | 33 | 61 (63 patients were randomised to the Isoflurane group, 2 of these did not receive treatment.)
Completed | 31 | 60
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Drug: Isoflurane: Volatile for sedation in the ICU
  Isoflurane: Inhalation vapour, liquid. Isoflurane delivered by the Sedaconda ACD-S device
- Total: Total of all reporting groups
Arm/Group | Drug: Midazolam | Drug: Isoflurane | Total
Number analyzed (Participants) | 33 | 61 | 94
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 28 | 47 | 75
  Adolescents (12-17 years) | 5 | 14 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 23 | 36
  Male | 20 | 38 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 23
  Not Hispanic or Latino | 13 | 28 | 41
  Unknown or Not Reported | 10 | 20 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 22 | 41 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 18 | 28
Weight [Mean (Standard Deviation); unit: kg] — Population: Data missing for 1 patient in the Isoflurane group. Safety set
  kg
    number analyzed (Participants) | 33 | 60 | 93
    (all) | 26.95 (19.68) | 28.83 (17.25) | 28.16 (18.06)
Height [Mean (Standard Deviation); unit: cm] — Population: Data missing from 3 patients in the Isoflurane group and from 1 patient in the Midazolam group. Safety set
  cm
    number analyzed (Participants) | 32 | 58 | 90
    (all) | 118.3 (21.5) | 125.8 (26.6) | 123.2 (25.1)
Height [Median (Full Range); unit: cm] — Population: Missing data for 3 patients in Isoflurane group and from 1 patient in Midazolam group. Safety set.
  cm
    number analyzed (Participants) | 32 | 58 | 90
    (all) | 112.5 [91 to 170] | 123.0 [90 to 185] | 117.0 [90 to 185]
Weight [Median (Full Range); unit: kg] — Population: Data missing for 1 patient in the Isoflurane group. Safety set
  kg
    number analyzed (Participants) | 33 | 60 | 93
    (all) | 21.60 [11.0 to 112.0] | 20.00 [11.8 to 90.0] | 20.00 [11.0 to 112.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time of Adequately Maintained Sedation Depth up to 48 Hours (± 6 Hours)
Description: Percentage of time of adequately maintained sedation within the COMFORT-B interval (light, moderate or deep sedation) prescribed at randomisation, monitored every 2 h for a minimum of 12 h (up to 48 h ± 6 h)
Time Frame: Minimum of 12 hours up to 48 hours (± 6 hours).
Population: Full Analysis set (FAS): The FAS included all randomised patients who received IMP and had at least a 6-hour sedation period and at least 3 blinded COMFORT-B-assessments. The FAS followed the intention-to-treat principle, i.e., patients were analysed according to the treatment group they were assigned to at randomisation. The main statistical analysis was performed on this population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 59
Percentage of time | 62.37 [44.70 to 80.04] | 68.94 [52.83 to 85.05]
Statistical Analysis 1: Comparison: Drug: Midazolam vs Drug: Isoflurane; Test type: Other — Least square means of the difference between the treatment groups, including a 2-sided 95% confidence interval was reported in the statistical analysis. The noninferiority criterion was a relative difference of less than 15% between treatment groups; Mixed Models Analysis — Noninferiority was defined as the entire 95% CI for the difference being above the noninferiority margin for the relative difference of -15%. Testing the hypothesis of no difference between isoflurane and midazolam; Least square means = 6.57, 95% CI 2-sided [-8.99 to 22.13]

2. Primary Outcome: Percentage of Time of Adequately Maintained Sedation Depth up to 48 Hours (± 6 Hours)
Description: as for outcome 1
Time Frame: Minimum of 12 hours up to 48 hours (± 6 hours).
Population: The PP analysis set included all patients in the FAS without any major protocol deviation affecting the primary analysis. To be included in the PP analysis patients had to have been sedated for at least 12h (which was interpreted as 12 h of study sedative treatment from start of IMP), with at least 50% of the planned COMFORT-B assessments performed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 29 | 56
Percentage of time | 65.57 [44.03 to 87.11] | 70.91 [50.75 to 91.07]
Statistical Analysis 1: Comparison: Drug: Midazolam vs Drug: Isoflurane; Test type: Non-Inferiority — The non-inferiority margin was set to a relative difference of -15%; Testing the hypothesis of no difference between isoflurane and midazolam; Least square means = 5.34, 95% CI 2-sided [-10.48 to 21.17]

3. Secondary Outcome: Compare the Use of Opioids
Description: Dose of opioids from first blinded COMFORT-B assessment (at +2 h from start of study drug) to end of study treatment period. This was a key secondary efficacy endpoint. Dose of opioids was expressed as fentanyl IV equivalents.
Time Frame: From first blinded COMFORT-B assessment (at +2 h from start of study drug initiation) to end of the study treatment period
Population: The FAS included all randomised patients who received IMP and had at least a 6-hour sedation period and at least 3 blinded COMFORT-B-assessments. The FAS followed the intention-to-treat (ITT) principle, i.e., patients were analysed according to the treatment group they were assigned to at randomisation.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/kg/h
Groups:
- Drug: Isoflurane: Volatile for sedation in the ICU
  Isoflurane: Inhalation vapour, liquid. Isoflurane delivered by the Sedaconda ACD-S.
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 59
μg/kg/h | 4.6 [3.5 to 5.6] | 2.1 [1.3 to 2.9]
Statistical Analysis 1: Comparison: Drug: Midazolam vs Drug: Isoflurane; Test type: Superiority; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.8 to -1.1]

4. Secondary Outcome: Compare the Use of Opioids
Description: Dose of opioids during the last 4 h of study treatment, as compared to the first 4 h of study treatment after first blinded COMFORT-B assessment. This was a key secondary efficacy endpoint. Dose of opioids is expressed as fentanyl IV equivalents.
Time Frame: Last 4 hours of study treatment compared to first 4 hours of study treatment after first blinded COMFORT-B assessment (at +2 h from start of study drug initiation).
Population: FAS: Patients with 8 hours or more of study treatment from first blinded COMFORT-B assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/kg/h
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 59
μg/kg/h | 0.58 [-0.16 to 1.32] | -0.19 [-0.74 to 0.35]
Statistical Analysis 1: Comparison: Drug: Midazolam vs Drug: Isoflurane; Test type: Superiority — Results display comparison between isoflurane and midazolam and are based on an analysis of variance model with treatment group as fixed effect and baseline opioid dose as covariate; p = 0.096, ANCOVA; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.69 to 0.14]

5. Secondary Outcome: Compare Time From End of Study Drug Administration to Extubation
Description: Time from end of study drug administration to extubation if study drug was terminated for extubation
Time Frame: From end of study drug administration to extubation or end of extubation attempt
Population: Subgroup of patients with endotracheal tube where wake-up was initiated at end of study treatment
Measure: Mean (Inter-Quartile Range); unit: hour
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 20 | 35
hour | 1.09 [0.49 to 5.50] | 0.75 [0.25 to 1.5]
Statistical Analysis 1: Comparison: Drug: Midazolam vs Drug: Isoflurane; Time to extubation; Test type: Superiority; p = 0.0021, Regression, Cox; Hazard Ratio (HR) = 3.3, 95% CI 2-sided [1.54 to 7.07]

6. Secondary Outcome: Compare the Proportion of Time With Spontaneous Breathing
Description: Proportion of observations with spontaneous breathing efforts during study treatment. This was a key secondary safety endpoint.
Time Frame: From initiation of study drug treatment to End of study treatment (up to 48h +/- 6h)
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of time
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 59
proportion of time | 0.44 [0.28 to 0.59] | 0.48 [0.36 to 0.60]
Statistical Analysis 1: Comparison: Drug: Midazolam vs Drug: Isoflurane; Spontaneous breathing efforts. Results display a comparison between isoflurane and midazolam and are based on a mixed effects analysis of variance model with treatment group as fixed effect; Test type: Superiority; p = 0.636, ANOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.15 to 0.25]

7. Secondary Outcome: Evaluate Haemodynamic Effect as Indicated by Need for Additional Inotropic/Vasopressor Agent
Description: Need for additional inotropic/vasopressor agent defined by change in Vasoactive-Inotropic Score (VIS) during study treatment period compared to baseline.
  The VIS quantifies the amount of cardiovascular support required by infants postoperatively according to the below calculation:
  VIS = dopamine (µg/kg/min) + dobutamine (µg/kg/min) + 100 × epinephrine (µg/kg/min) + 100 × norepinephrine (µg/kg/min) + 10 × milrinone (µg/kg/min) + 10,000 × vasopressin (U/kg/min).
  An increased VIS score correlates to an increase in inotropic/vasopressor agents.
Time Frame: From start of study treatment to end of study treatment (up to 48h +/- 6h)
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Change from baseline in VIS
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 61
Change from baseline in VIS
  ≤24 hours | 5.4 (19.3) | 3.4 (19.9)
  >24 hours | 1.9 (9.7) | 8.8 (44.4)
Statistical Analysis 1: Comparison: Drug: Midazolam vs Drug: Isoflurane; Need for inotropic/vasopressor agent at ≤24 hours; Test type: Superiority — Results display comparison between isoflurane and midazolam and are based on a Wilcoxon ranksum test; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Drug: Midazolam vs Drug: Isoflurane; Need for inotropic/vasopressor agent at >24 hours; Test type: Superiority; p = 0.637, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Evaluate the Number of Patients With Withdrawal Symptom
Description: Evaluate the frequency of withdrawal symptoms in isoflurane- vs midazolam-treated patients according to SOS-PD.
Time Frame: From > 96 hours sedation (including pre-study sedation period) until the end of the 48-hour post study treatment monitoring or ICU discharge, whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 61
Participants | 2 | 3

9. Secondary Outcome: Evaluate the Frequency of Delirium
Description: Evaluate the frequency of delirium in isoflurane- vs midazolam-treated patients
Time Frame: Patients admitted to the ICU ≥48 hours (including period prior to study enrolment) until the end of the 48-hour post study treatment monitoring or ICU discharge, whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 61
Participants | 5 | 12

10. Secondary Outcome: Evaluate the Frequency of Neurological Symptoms or Psychomotor Dysfunction
Description: Evaluate the frequency of neurological symptoms or psychomotor dysfunction during and up to 48 hours after discontinuation of isoflurane and midazolam treatment, and the association with duration of treatment, and total exposure (MAC hours and midazolam doses) over time.
Time Frame: During study treatment and up to 48 hours after discontinuation of isoflurane and midazolam
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 61
Participants | 6 | 16

11. Secondary Outcome: Compare the 30 Days/Hospital Mortality
Description: Compare the 30 days/hospital mortality in isoflurane- vs midazolam-treated patients
Time Frame: From start of study treatment up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 61
Participants | 2 | 0

12. Secondary Outcome: Compare Ventilator-free Days
Description: Ventilator-free days at 30 days from start of study treatment period.
Time Frame: From start of study treatment up to 30 days
Population: Safety analysis set (only patients not withdrawn prior to day 30)
Measure: Mean (Standard Deviation); unit: Number of ventilator-free days
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 60
Number of ventilator-free days | 22.55 (10.62) | 25.00 (6.74)

13. Secondary Outcome: Compare the Time in ICU/Hospital
Description: Compare the time in ICU at 30 days from start of study treatment period. This was a secondary safety endpoint. Patients that were withdrawn prior to day 30 were excluded from the analysis. Patients who died before day 30 were not considered withdrawals. For these patients, the days in ICU until day of death were considered ICU days.
Time Frame: From start of study treatment up to 30 days
Population: Safety analysis set (only patients not withdrawn prior to day 30)
Measure: Mean (Standard Deviation); unit: Number of ICU days
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 60
Number of ICU days | 10.21 (9.13) | 9.65 (7.87)

14. Secondary Outcome: Compare ICU-free Days
Description: Compare ICU-free days up to 30 days in isoflurane- vs midazolam-treated patients.
Time Frame: From start of study treatment up to 30 days
Population: Safety analysis set (only patients not withdrawn prior to day 30). This was a secondary safety endpoint. Patients who died before day 30 were not considered withdrawals. For these patients, the days in ICU until day of death were considered ICU days.
Measure: Mean (Standard Deviation); unit: Number of days alive and not in the ICU
Arm/Group | Drug: Midazolam | Drug: Isoflurane
Number analyzed (Participants) | 33 | 60
Number of days alive and not in the ICU | 18.58 (10.26) | 20.35 (7.87)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded during the study drug treatment period (up to 48h +/- 6h from start of IMP) and for 48 hours after end of study drug treatment. Mortality was monitored for up to 30 days.
Arm/Group | Drug: Midazolam | Drug: Isoflurane
All-Cause Mortality (participants affected / at risk) | 2/33 | 1/61
Serious Adverse Events (participants affected / at risk) | 8/33 | 19/61
Other Adverse Events (participants affected / at risk) | 13/33 | 32/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Midazolam (N=33) | Drug: Isoflurane (N=61)
Magnetic resonance imaging head abnormal (Investigations) | 0 (0) | 1 (1)
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complications of transplanted liver subjects affected / exposed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Postoperative wound infection (General disorders) | 0 (0) | 1 (1)
Pseudomembranous colitis (General disorders) | 1 (1) | 0 (0)
Pyelonephritis (General disorders) | 0 (0) | 1 (1)
Septic shock (General disorders) | 2 (2) | 0 (0)
Urinary tract infection (General disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Midazolam (N=33) | Drug: Isoflurane (N=61)
Hyperthermia (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 8 (13)
Hypoxia (General disorders) | 1 (3) | 4 (12)
Pleural effusion (General disorders) | 1 (2) | 5 (6)
Delirium (Psychiatric disorders) | 1 (1) | 5 (5)
Bradycardia (Cardiac disorders) | 3 (10) | 3 (12)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (8)
Constipation (Gastrointestinal disorders) | 4 (4) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT04684238/Prot_SAP_000.pdf